CLINICAL TRIAL: NCT02289300
Title: A Phase II Randomized, Double-Blind, Placebo Controlled, Parallel Study of DCB-BO1202 for Alleviating Liver Fibrosis in HBV Patients With Intermediate Hepatocellular Carcinoma Receiving Loco-regional Therapies
Brief Title: A Study to Evaluate a Study Drug, DCB-BO1202, for Alleviating Liver Fibrosis in Liver Cancer Patients
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: At sponsor's discretion
Sponsor: A2 Healthcare Taiwan Corporation (Industry)
Collaborators: GoldenMed BioTechnology (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BO1202-LF1201
Record Dates: First submitted 2014-11-07; First posted 2014-11-13 (Estimated); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Liver Fibrosis; HEPATITIS B CHRONIC; Hepatocellular Carcinoma
MeSH Terms: conditions — Liver Cirrhosis; Hepatitis B, Chronic; Carcinoma, Hepatocellular

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- DCB-BO1202 (Experimental)
  Interventions: Drug: DCB-BO1202
- DCB-BO1202+Placebo (Experimental)
  Interventions: Drug: DCB-BO1202+Placebo
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DCB-BO1202 — The assignment will be as follows:
  (Each DCB-BO1202 300mg capsule contains 150mg active ingredient)
  DCB-BO1202: 4 DCB-BO1202 300mg capsules, t.i.d., orally.
  Duration of Administration: 96 weeks ((11 treatment weeks + 1 observation week) * 8 cycles)
  Arms: DCB-BO1202
Drug: Placebo — The assignment will be as follows:
  Placebo: 4 matched placebo, t.i.d., orally.
  Duration of Administration: 96 weeks ((11 treatment weeks + 1 observation week) * 8 cycles)
  Arms: Placebo
Drug: DCB-BO1202+Placebo — The assignment will be as follows:
  (Each DCB-BO1202 300mg capsule contains 150mg active ingredient)
  DCB-BO1202+Placebo: 2 DCB-BO1202 300mg capsules plus 2 matched placebo, t.i.d., orally.
  Duration of Administration: 96 weeks ((11 treatment weeks + 1 observation week) * 8 cycles)
  Arms: DCB-BO1202+Placebo

SUMMARY:
The purpose of this study is to determine whether an investigational drug DCB-BO1202 is effective and safe in the treatment of liver fibrosis in HBV patients having experienced intermediate stage hepatocellular carcinoma (HCC)

DETAILED DESCRIPTION:
The study will include the first 188 subjects who are randomized. The purpose of study is to collect efficacy results to evaluate treatment effect on the primary endpoint. The second endpoints is to evaluate drug safety on the incidence of the primary endpoint through the treatment period.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 20-65 years (inclusive) of either gender
2. With evidence of HBV infection confirmed by positive for Hepatitis B virus antigen (HBsAg)
3. With Barcelona Clinic Liver Cancer (BCLC) intermediate stage (BCLC-B) hepatocellular carcinoma (HCC)
4. Having received radiofrequency ablation (RFA) or transarterial embolization (TAE) for hepatitis B virus (HBV) related hepatocellular carcinoma at least 4 weeks before Screening
5. With liver stiffness measurement (assessed by Fibroscan®) of 7-20 kPa
6. Able to understand and willing to sign the informed consent

Exclusion Criteria:

1. Evidence or history of chronic hepatitis caused by Hepatitis C virus (HCV)
2. With abnormal organ functions such as absolute neutrophil count (ANC) < 1500 /μL, hemoglobin < 9 gm/dL, platelets < 50,000 /μL, creatinine > 2 mg/dL, alanine aminotransferase (AST) or ALT > 5 X upper normal limit of the current institution; bilirubin > 2.5 mg/dL, prothrombin time (PT) prolongation > 4 sec above upper limit of normal
3. With uncontrolled infection or serious infection within the past 4 weeks
4. With any other carcinoma except skin cancer
5. Women who are pregnant or breast-feeding or with child-bearing potential but unable or unwilling to practice a highly effective means of contraception
6. Active substance abuse, including alcohol, which, in the opinion of the investigator, risks impairing the ability of the patient to comply with the protocol
7. History of allergy to any substance of investigational products
8. With known human immunodeficiency virus (HIV) infection
9. Judged to be not applicable to this study by investigator such as difficulty of follow-up observation
10. With any other serious diseases/medical history considered by the investigator not in the condition to enter the trial
11. Administered with any anti-HBV drugs within 4 weeks of entering this study. (Note: Anti-HBV treatments are allowed to be taken during study period when necessary.)
12. Having participated other investigational study within 4 weeks of entering this study

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-01 (Estimated); Primary Completion 2021-01 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in liver stiffness measurement (kPa) assessed by Fibroscan® at Final visit | 96 weeks

SECONDARY OUTCOMES:
Change from baseline in liver stiffness measurement (kPa) assessed by (Fibroscan®) at each post-treatment visit | Weeks 4, 8, 12, 24, 36, 48, 60, 72, 84
Changes from baseline in biomarkers associated with liver fibrosis at each post-treatment visit compared to baseline | Weeks 4, 8, 12, 24, 36, 48, 60, 72, 84, 96
Changes from baseline in hepatic functions such as liver enzymes, albumin, direct bilirubin and international normalize ratio (INR) at each post-treatment visit compared to baseline | Weeks 4, 8, 12, 24, 36, 48, 60, 72, 84, 96
Change from baseline in log10 HBV deoxyribonucleic acid (DNA) measured by Polymerase chain reaction (PCR) assay at each post-treatment visit and each of post-study follow-up visits compared to baseline | Weeks 4, 8, 12, 24, 36, 48, 60, 72, 84, 96
Transition of HBV DNA detectable status (e.g. <500 copies/mL) by PCR at each post-treatment visit from baseline | Weeks 4, 8, 12, 24, 36, 48, 60, 72, 84, 96
Change in Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue total score and sub-scores compared to baseline at each post-treatment visit | Weeks 4, 8, 12, 24, 36, 48, 60, 72, 84, 96
Overall survival rates at Week-48 and Week-96 visits | Weeks 48, 96
Recurrence rate at Week-96 visit | Week 96
Time to recurrence of cancer | Weeks 4, 8, 12, 24, 36, 48, 60, 72, 84, 96
Incidence of adverse events (AEs) | Weeks 4, 8, 12, 24, 36, 48, 60, 72, 84, 96
Changes from baseline to post-treatment visits in vital signs, laboratory examination, and physical examinations results | Weeks 4, 8, 12, 24, 36, 48, 60, 72, 84, 96

CONTACTS AND LOCATIONS:
Overall Officials: Kai-Wen Huang, MD, Principal Investigator — Hepatitis Research Center, Department of Surgery, National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan